CLINICAL TRIAL: NCT04867200
Title: An Open Label, Randomized, Single-dose, 2-sequence, 2-period, Cross-over Phase 1 Study to Evaluate the Safety and Pharmacokinetics of CKD-344 in Healthy Adult Volunteers
Brief Title: A Clinical Study to Evaluate the Safety and Pharmacokinetics of CKD-344 in Healthy Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A109_02BE2106
Record Dates: First submitted 2021-04-27; First posted 2021-04-30 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Anticoagulant
MeSH Terms: interventions — Drug Evaluation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): 1. Period 1: Reference drug(Lixiana 60 mg)
  2. Period 2: Test drug(CKD-344 60 mg)
  Interventions: Drug: Lixiana(D006); Drug: CKD-344
- Group B (Experimental): 1. Period 1: Test drug(CKD-344 60 mg)
  2. Period 2: Reference drug(Lixiana 60 mg)
  Interventions: Drug: Lixiana(D006); Drug: CKD-344

INTERVENTIONS:
Drug: Lixiana(D006) — NOAC(Factor Xa inhibitor)
  Other Names: Reference Drug
Drug: CKD-344 — NOAC(Factor Xa inhibitor)
  Other Names: Test Drug

SUMMARY:
A Clinical Trial to evaluate the Pharmacokinetics and safety of CKD-344

DETAILED DESCRIPTION:
A Phase 1 Clinical Trial to evaluate the safety and pharmacokinetics in healthy adult volunteers after administration of CKD-344.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult volunteers aged ≥ 19 years
2. Weight ≥60kg, with calculated body mass index(BMI) of 18 to 30 kg/m2
3. Those who have no congenital diseases or chronic diseases and have no abnormal symptoms or findings.
4. Those who are eligible for clinical trials based on laboratory (hematology, blood coagulation, blood chemistry, serology, urinalysis) at screening.
5. Those who agree to contraception during the participation of clinical trial.
6. Those who voluntarily decide to participate and agree to comply with the cautions after fully understand the detailed description of this clinical trial.

Exclusion Criteria:

1. Those who has a medical evidence or a history of clinically significant gastrointestinal, cardiovascular, endocrine, pulmonary, hematological, infective disease, renal, urinary, psychiatric, neurologic, skeletomuscular, immune, etc.
2. Those who have a history of gastrointestinal surgery except simple appendectomy and hernia surgery.
3. Those who had taken prescription or nonprescription drugs within 10 days prior to the first dose of investigational product.
4. Those who received investigational products or participated in bioequivalence tests within 6 months before the first administration of clinical trial drugs.
5. Those who donated whole blood within 8 weeks or blood components within 4 weeks prior to the first dose of the investigational product.
6. Those who exceed an alcohol and cigarette consumption than below criteria. A. Alcohol: Man- 21 glasses/week, Woman - 14 glasses/week B. Smoking: 20 cigarettes/day
7. Those who exceeds 2 times the upper limit of the reference range of AST(or ALT) or 1.5 times the upper limit of the reference range of γ-GTP.
8. Those who have hypersensitivity to the drug or the drug ingredient, such as anaphylactic reactions.
9. Those who have specific disease(e.g. severe bleeding disorder, severe renal/hepatic disease, uncontrolled severe hypertension, etc.)
10. Those who were deemed inappropriate to participate in the study by the investigator.
11. Those who have a pregnant or nursing woman.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-04-27 (Actual); Primary Completion 2021-05-25 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
AUCt(Area Under Curve last) of CKD-344 | predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 hours post-dose
  Area under the plasma concentration time curve of CKD-344, from time zero up to the last measurable concentration.
Cmax | predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 hours post-dose
  The maximum concentration observed of CKD-344 over blood sampling time.

CONTACTS AND LOCATIONS:
Overall Officials: Yook-Hwan Noh, Principal Investigator — South Korea
Locations (1):
- H+ Yangji Hospital, Seoul, South Korea